CLINICAL TRIAL: NCT01403233
Title: An Open-label, Sequential Supplementation Study Comparing the Bioavailability of Two Doses of cogniVida™ With One Dose of Rebaudioside A in Healthy Male Subjects
Brief Title: Bioavailability of Two Doses of cogniVida™ With One Dose of Rebaudioside A in Healthy Male Subjects
Acronym: StevReb-PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-06-01-STEV
Record Dates: First submitted 2011-07-19; First posted 2011-07-27 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety
MeSH Terms: interventions — rebaudioside A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cogniVida™ 50 mg/day (Experimental)
  Interventions: Dietary Supplement: cogniVida 50mg/day
- cogniVida™ 100 mg/day (Experimental)
  Interventions: Dietary Supplement: cogniVida100mg/day
- Rebaudioside-A 303.7 mg/day (Active Comparator)
  Interventions: Dietary Supplement: Rebaudioside-A 303.7mg/day

INTERVENTIONS:
Dietary Supplement: cogniVida 50mg/day — 2 capsules 25 mg (total 50 mg) cogniVida™ once a day
  Arms: cogniVida™ 50 mg/day
Dietary Supplement: cogniVida100mg/day — 4 capsules 25 mg (total 100 mg) cogniVida™ once a day
  Arms: cogniVida™ 100 mg/day
Dietary Supplement: Rebaudioside-A 303.7mg/day — 4 capsules 75.92 mg (total 303.68 mg) rebaudioside A once a day
  Arms: Rebaudioside-A 303.7 mg/day

SUMMARY:
The purpose of the study is to examine the bioavailability of cogniVida™ in 10 healthy male subjects after consumption of two different doses of cogniVida™ (50 mg and 100 mg) and to compare the plasma values with values obtained in subjects receiving rebaudioside A (303.68 mg). In addition, also safety and tolerability parameters 24 hours after ingestion of the study compounds will be determined.

cogniVida™ is considered a dietary supplement, and therefore it is not an approved drug by the Food and Drug Administration (FDA). It is regulated like a food. The U.S. Food and Drug Administration does not strictly regulate herbs and dietary supplements. The investigators do not claim that this supplement is meant to treat any ailment.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male, age 30 - 50 years
* Subject is willing to maintain his or her habitual diet and physical activity patterns throughout the study period.
* Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results
* Subject has a body mass index (BMI) of ≥20.00 and <28.00 kg/m2 at screening.
* Subject is willing to refrain from consuming drinks containing grapefruit 7 days prior to test days.
* Subject is willing to refrain from consuming caffeine, caffeine-containing products and alcoholic drinks 24 h prior to test days and until the end of each assessment period.
* Subject is willing to refrain from vigorous physical activity 12 h prior to test days.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subject has a positive drug screening of amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, 3,4-methylenedioxymethamphetamine, opiates or tricyclic antidepressants at screening.
* Subjects has a positive blood alcohol and breath carbon monoxide test at screening.
* Subject has abnormal laboratory test results of clinical significance, including, but not limited to: Epidermal-Growth-Factor-Receptor (eGFR) <60mL/min/1.73m2, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥1.5X the upper limit of normal at screening.
* Subject has donated more than 300 mL of blood or has lost a significant amount of blood during the three months prior to screening.
* Anemia of any etiology defined as hemoglobin < 140g/L for males and < 123g/L for female
* Subject has uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the average blood pressure measured at screening.
* Subject has a history or presence of cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorders.
* Subject has a history, in the judgment of the Investigator, of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Subject has a history or presence of cancer in the prior five years, except for non-melanoma skin cancer.
* Excessive habitual caffeine consumption (>300 mg caffeine/d or ≥ 3 cups of caffeinated coffee/d), following screening and throughout the study period.
* Use of antibiotics or signs of active systemic infection. Treatment visits will be rescheduled to allow the subject to wash off of the antibiotic for at least one month prior to any test visit.
* Use of dietary supplements containing any of the following: ginkgo biloba, St. John's wort, ginseng, gotu kola (Indian pennywort); daily doses of vitamin E (≥30 mg/d) or folic acid (≥400 ug/d); thiamine, riboflavin, and/or pyridoxine (≥2 mg/d); and eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA)or a combination of EPA + DHA (≥500 mg/d) within 2 weeks prior to screening.
* Consumption of stevia extract (reb A / steviosides) sweetened products/drinks or stevia leaves within one month of the study.
* Subject has had exposure to any non-registered drug product within 30 days prior to the screening visit.
* Recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Subject has a known allergy or sensitivity to study product or any ingredients of the study product or meals provided.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma Area under the Curve (AUC) (0-72 hours) being produced after cogniVida™ (50 and 100 mg) and rebaudioside A (303.68 mg) consumption | 0 - 72 hours
  Blood sampling timepoints: cogniVida: 0 min, 15min, 30min, 45min, 1h, 1:30h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 48, and 72h after dosing.
  RebA: 0 min, 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36, 48, and 72h after dosing

SECONDARY OUTCOMES:
Time to plasma peak (Tmax) being produced after cogniVida™ (50 and 100 mg) and rebaudioside A (303.68 mg) consumption | 0 - 72 hours
  Blood sampling timepoints: cogniVida: 0 min, 15min, 30min, 45min, 1h, 1:30h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 48, and 72h after dosing.
  RebA: 0 min, 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36, 48, and 72h after dosing
Plasma Peak Concentration (Cmax) being produced after cogniVida™ (50 and 100 mg) and rebaudioside A (303.68 mg) consumption | 0 - 72 hours
  Blood sampling timepoints: cogniVida: 0 min, 15min, 30min, 45min, 1h, 1:30h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 48, and 72h after dosing.
  RebA: 0 min, 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36, 48, and 72h after dosing
Time to reach half of peak concentration in plasma T1/2 being produced after cogniVida™ (50 and 100 mg) and rebaudioside A (303.68 mg) consumption | 0 - 72 hours
  Blood sampling timepoints: cogniVida: 0 min, 15min, 30min, 45min, 1h, 1:30h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 48, and 72h after dosing.
  RebA: 0 min, 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36, 48, and 72h after dosing
Vital signs | 24 hours after each supplementation
  Vital signs as safety parameters being measured 24 h after each supplementation.
White blood cell (WBC) count (Routine Haematology) | 24 hours after each supplementation
  White blood cells will be counted as a routine haematology parameter to assess safety 24 h after each supplementation.
Hemoglobin (Routine Haematology) | 24 hours after each supplementation
  Hemoglobin will be measured as a routine haematology parameter to assess safety 24 h after each supplementation.
Blood urea nitrogen (BUN) (Clinical Chemistry) | 24 hours after each supplementation
  Blood urea nitrogen will be measured as a routine clinical chemistry parameter to assess safety 24 h after each supplementation.
Cystatin-C (Clinical Chemistry) | 24 hours after each supplementation
  Cystatin-C will be measured as a routine clinical chemistry parameter to assess safety 24 h after each supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc, London, Ontario, Canada